CLINICAL TRIAL: NCT00379444
Title: Tobacco Cessation Treatment for Pregnant Alaska Natives
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1711-05; 5R01DA025156-03 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2006-09

CONDITIONS: Tobacco Use
Keywords: tobacco, intervention, tobacco cessation, ALaska Natives,; Native Americans, pregnancy, women
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation | interventions — Counseling; S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Standard intervention (counseling + self-help written materials) — counseling
Behavioral: Enhanced Intervention (same as standard treatment plus 10-15 min of counseling and a culturally tailored video) — counseling

SUMMARY:
This study will develop a culturally appropriate tobacco cessation behavioral intervention for Alaska Native women who are pregnant and who use tobacco. We will examine the feasibility of the intervention in terms of recruitment and retention of participants, acceptability to patients and prenatal health care providers, and the potential effectiveness of the tobacco use intervention.

DETAILED DESCRIPTION:
Tobacco use is the single largest cause of premature and preventable death in the U.S. The prevalence of tobacco use among adults is currently highest among Alaska Natives. Over 50% of Alaska Native women residing in the Yukon-Kuskokwim (Y-K) Delta of western Alaska use smokeless tobacco or smoke cigarettes during pregnancy. Alaska Natives of this region are of Yup'ik or Cup'ik Eskimo, or Athabascan Indian ethnicity. No prior work has evaluated tobacco use interventions for pregnant Alaska Native women.

This proposal builds on our successful partnership and track record of collaboration with Y-K Delta Alaska Natives. The objective of this R21 proposal is to develop and pilot test a novel, culturally-tailored behavioral approach to tobacco cessation for pregnant Alaska Native women. We expect that as a result of this project, we will have developed a replicable, feasible, and acceptable counseling intervention, the efficacy of which can be tested in future larger-scale randomized clinical trials. Social cognitive (learning) theory is the conceptual basis for the proposed intervention.

This project will take place in two phases. In Phase 1, we will develop a multi-component, culturally-tailored, tobacco use intervention with and for Alaska Native pregnant women, including a videotape and telephone counseling. This work will include development of a counselor manual and development of the intervention with focus groups. During this phase, 10 pregnant women will complete the protocol, which will be modified and refined based on feedback from participants and counselors. Phase 2, consisting of a pilot clinical trial, will apply a randomized, two group design with assessments at the first prenatal visit (baseline) and at the last prenatal visit approximately 36 weeks gestation. Pregnant women will be recruited and randomized to either a standard (N=30) or enhanced (N=30) tobacco use intervention. The overall health related objective of this line of research is to develop effective treatment programs with and for Alaska Native pregnant women that will ultimately reduce the risk of tobacco-related disease.

ELIGIBILITY:
Inclusion Criteria:

For pilot testing of the intervention, we will recruit 70 Alaska Native adult pregnant women (10 in Phase 1, 60 in Phase 2) at their first prenatal visit. To be eligible, the participant must: (1) be 18 years of age or older, (2) provide written informed consent, (3) be willing and able to participate in all aspects of the study, (4) be <24 weeks pregnant, (4) self-report any use of Iqmik, commercial ST, and/or cigarette smoking during the past 7 days, (5) plan to make a serious attempt to stop tobacco use within the next 30 days, (6) have access to a working telephone or provide phone number of a family member, and (7) have access to a working television and VCR in the home or other location.

Exclusion Criteria:

Women will be excluded if: (1) they are currently (past 30 days) participating in any tobacco treatment or (2) if there is another study participant from the same household.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Tobacco abstinence, feasibility (recruitment and retention), | end of pregnancy
acceptability of the intervention to the women and providers. | week 6

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, P, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States